CLINICAL TRIAL: NCT05870345
Title: The Diagnostic Accuracy of Pocket Size Ultrasound (PsUS) in the Detection of Pediatric Elbow Fractures
Brief Title: Pocket Sized Ultrasound (PsUS) and Pediatric Elbow Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB21-0678
Record Dates: First submitted 2023-04-04; First posted 2023-05-23 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Elbow Injury; Elbow Fracture
Keywords: Pocket sized ultrasound; Pediatric elbow injury; Pediatric elbow fracture
MeSH Terms: conditions — Elbow Injuries; Elbow Fractures

STUDY DESIGN:
Intervention Model Description: Each participant receives the study intervention which is a pocket-sized ultrasound exam.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ultrasound Exam (Other): The Study consists of two parts, a feasibility part and an active part.
  Participants in the feasibility part of the study only undergo a pocket-sized ultrasound exam and are distinct (unique) group with no overlap or involvement with the active part.
  Participants in the active part of the study undergo a pocket-sized ultrasound exam and continue with normal clinically indicated medical care in the ED. The comparison to the ultrasound images is either a X-ray if fracture is suspected or bedside nursemaid reduction if subluxation is suspected (participants will act as their own comparison based on their routine ED clinical management). There is no participation overlap with the feasibility part.
  Interventions: Device: Butterfly IQ

INTERVENTIONS:
Device: Butterfly IQ — Butterfly IQ is a pocket sized ultrasound device. Each participant will undergo a ultrasound exam of both elbows using a pocket sized ultrasound device.

SUMMARY:
The main purpose of this project is to investigate the accuracy of pocket-sized ultrasound (PsUS) in the diagnosis of pediatric elbow fractures. The primary research objective is to determine the test performance characteristics of PSUS performed by pediatric emergency medicine physicians compared to radiography for the detection of pediatric elbow fractures. The project will consist of two parts, first involving a feasibility study and followed by an active study. The feasibility study will aim to answer if providers can perform an adequate elbow ultrasound exam after a brief study training. The active study will investigate the initial accuracy of the PsUS. Participants will be asked in either the feasibility or the active phases of the study to undergo a brief pocket-sized ultrasound elbow exam of both elbows. Patient will continue to receive their previously determined clinical ED management. In the active phase of the study, participant's elbow X-rays or if patient underwent bedside nursemaid reduction will be the comparison to pocket-sized ultrasound images.

DETAILED DESCRIPTION:
The main purpose of this project is to investigate the accuracy of pocket-sized ultrasound (PsUS) in the diagnosis of pediatric elbow fractures. The primary research objective is to determine the test performance characteristics of PSUS performed by pediatric emergency medicine physicians compared to radiography for the detection of pediatric elbow fractures. The project will consist of two parts, first involving a feasibility study and followed by an active study.

This project will consist of two parts, involving first a brief feasibility phase followed by a pilot study conducted in an urban pediatric emergency department (Comer Children's Hospital in Chicago, IL). For the feasibility phase, the purpose is to demonstrate that novice PsUS users are able to obtain accurate and adequate imaging for interpretation. This phase will initially involve the study providers receiving the elbow PsUS exam training. Once trained, each study provider will obtain 3 elbow exams of participants between the ages of 1-16 years old. Providers will use the standardized views reviewed in the ultrasound training to perform the exam, with verbal consent obtained from each participant's parent for inclusion in the feasibility study. These images will be reviewed by study staff to ensure US examiners are obtaining the correct standardized views.

Once the feasibility exams are completed, the study providers are able to begin active study recruitment which will involve recruiting children between the ages of 1-16 years old with isolated acute elbow pain. Parents will initially be approached in the emergency department (ED), with written consent obtained if interested and eligible. Once consented, patients will undergo bilaterally standardized elbow exams using the pocket-sized ultrasound. All images will be stored on a password protected, cloud-based imaging database with all identifying information removed. After the exam, a basic assessment of the images will be made by the bedside ultrasound provider, as positive, negative or equivocal for signs of elbow fracture, but before reviewing any radiographic imaging. A positive PsUS will be defined as the presence of signs of elbow fracture, either as direct signs including cortical discontinuities or indirect signs including posterior fat pad with or without lipohemarthrosis on ultrasound exam. Following the ultrasound exam, patients will undergo standard clinical care for acute elbow injury per primary ED team which may consist of Xray or possible bedside nursemaid reduction. When applicable, study investigators will review the final blinded radiology readings of the initial or subsequent x-ray images after the patient encounter. Additionally, research staff will also attempt to follow up with participants after their ED visit for their elbow injury to determine if any additional radiographic imaging or care was obtained and if subsequent occult fractures were discovered on later imaging that may have been missed on the initial evaluation.

The primary aim of the feasibility portion of the study is to determine acceptability of the PsUS study training to obtain adequate elbow images. The primary aim of the active study is to compare the initial test performance characteristics of PSUS performed by bedside physicians compared to standard radiography in the diagnosis of pediatric elbow fractures.

ELIGIBILITY:
Inclusion Criteria:

For Feasibility phase: children between the ages of 1-16 years olds

For Active phase: children between the ages of 1-16 years olds with isolated, acute (less than 48 hrs) elbow pain in the setting of adequate history of trauma

Exclusion Criteria:

Both phases:

* Children <1 or >16 years old
* Those with open fractures, gross deformities, multiple traumatic injuries, distal neurovascular compromise, unstable vital signs or hemodynamic instability, altered mental status, history of skeletal abnormalities, or past elbow fracture as well as wards of the state or those unable to provide consent
* Patients who have a confirmed diagnosis of fracture at an outside institutions prior to arrival to the ED will also be excluded

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Benjamin, MD, Principal Investigator — University of Chicago/Comer Children's Hospital
Locations (1):
- University of Chicago/Comer Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share information with other researchers

REFERENCES:
- [Background] Tsou PY, Ma YK, Wang YH, Gillon JT, Rafael J, Deanehan JK. Diagnostic accuracy of ultrasound for upper extremity fractures in children: A systematic review and meta-analysis. Am J Emerg Med. 2021 Jun;44:383-394. doi: 10.1016/j.ajem.2020.04.071. Epub 2020 Apr 27. PMID 32507477
- [Background] Lee SH, Yun SJ. Diagnostic Performance of Ultrasonography for Detection of Pediatric Elbow Fracture: A Meta-analysis. Ann Emerg Med. 2019 Oct;74(4):493-502. doi: 10.1016/j.annemergmed.2019.03.009. Epub 2019 May 9. PMID 31080032
- [Background] Ackermann O, Liedgens P, Eckert K, Chelangattucherry E, Ruelander C, Emmanouilidis I, Ruchholtz S. Ultrasound diagnosis of juvenile forearm fractures. J Med Ultrason (2001). 2010 Jul;37(3):123-7. doi: 10.1007/s10396-010-0263-x. Epub 2010 Apr 23. PMID 27278011
- [Background] Ackermann O, Simanowski J, Eckert K. Fracture Ultrasound of the Extremities. Ultraschall Med. 2020 Feb;41(1):12-28. doi: 10.1055/a-1023-1782. Epub 2020 Feb 5. PMID 32023628
- [Background] Eckert K, Ackermann O, Schweiger B, Radeloff E, Liedgens P. Ultrasound evaluation of elbow fractures in children. J Med Ultrason (2001). 2013 Oct;40(4):443-51. doi: 10.1007/s10396-013-0446-3. Epub 2013 Apr 16. PMID 27277459
- [Background] Rabiner JE, Khine H, Avner JR, Friedman LM, Tsung JW. Accuracy of point-of-care ultrasonography for diagnosis of elbow fractures in children. Ann Emerg Med. 2013 Jan;61(1):9-17. doi: 10.1016/j.annemergmed.2012.07.112. Epub 2012 Nov 9. PMID 23142008
- [Background] McNeil CR, McManus J, Mehta S. The accuracy of portable ultrasonography to diagnose fractures in an austere environment. Prehosp Emerg Care. 2009 Jan-Mar;13(1):50-2. doi: 10.1080/10903120802474513. PMID 19145524
- [Background] Lau BC, Robertson A, Motamedi D, Lee N. The Validity and Reliability of a Pocket-Sized Ultrasound to Diagnose Distal Radius Fracture and Assess Quality of Closed Reduction. J Hand Surg Am. 2017 Jun;42(6):420-427. doi: 10.1016/j.jhsa.2017.03.012. Epub 2017 Apr 29. PMID 28460717
- [Background] Burnier M, Buisson G, Ricard A, Cunin V, Pracros JP, Chotel F. Diagnostic value of ultrasonography in elbow trauma in children: Prospective study of 34 cases. Orthop Traumatol Surg Res. 2016 Nov;102(7):839-843. doi: 10.1016/j.otsr.2016.07.009. Epub 2016 Sep 30. PMID 27697406
- [Background] Rennie L, Court-Brown CM, Mok JY, Beattie TF. The epidemiology of fractures in children. Injury. 2007 Aug;38(8):913-22. doi: 10.1016/j.injury.2007.01.036. Epub 2007 Jul 12. PMID 17628559
- [Background] Poonai N, Myslik F, Joubert G, Fan J, Misir A, Istasy V, Columbus M, Soegtrop R, Goldfarb A, Thompson D, Dubrovsky AS. Point-of-care Ultrasound for Nonangulated Distal Forearm Fractures in Children: Test Performance Characteristics and Patient-centered Outcomes. Acad Emerg Med. 2017 May;24(5):607-616. doi: 10.1111/acem.13146. Epub 2017 Apr 27. PMID 27976448
- [Background] Lee A, Colen DL, Fox JP, Chang B, Lin IC. Pediatric Hand and Upper Extremity Injuries Presenting to Emergency Departments in the United States: Epidemiology and Health Care-Associated Costs. Hand (N Y). 2021 Jul;16(4):519-527. doi: 10.1177/1558944719866884. Epub 2019 Aug 23. PMID 31441332
- [Background] Naranje SM, Erali RA, Warner WC Jr, Sawyer JR, Kelly DM. Epidemiology of Pediatric Fractures Presenting to Emergency Departments in the United States. J Pediatr Orthop. 2016 Jun;36(4):e45-8. doi: 10.1097/BPO.0000000000000595. PMID 26177059
- [Background] Bellavia MA, Cambise C, Coraci D, Maccauro G, Valassina A, Padua L. Ultrasound is a useful tool to evaluate nerve involvement in children with supracondylar humerus fractures. Muscle Nerve. 2017 Sep;56(3):E18-E20. doi: 10.1002/mus.25636. Epub 2017 Jun 5. No abstract available. PMID 28249353
- [Background] Chaar-Alvarez FM, Warkentine F, Cross K, Herr S, Paul RI. Bedside ultrasound diagnosis of nonangulated distal forearm fractures in the pediatric emergency department. Pediatr Emerg Care. 2011 Nov;27(11):1027-32. doi: 10.1097/PEC.0b013e318235e228. PMID 22068062
- [Background] Chen L, Baker MD. Novel applications of ultrasound in pediatric emergency medicine. Pediatr Emerg Care. 2007 Feb;23(2):115-23; quiz 124-6. doi: 10.1097/PEC.0b013e3180302c59. PMID 17351413
- [Background] Barata I, Spencer R, Suppiah A, Raio C, Ward MF, Sama A. Emergency ultrasound in the detection of pediatric long-bone fractures. Pediatr Emerg Care. 2012 Nov;28(11):1154-7. doi: 10.1097/PEC.0b013e3182716fb7. PMID 23114237
- [Background] Cho KH, Lee SM, Lee YH, Suh KJ. Ultrasound diagnosis of either an occult or missed fracture of an extremity in pediatric-aged children. Korean J Radiol. 2010 Jan-Feb;11(1):84-94. doi: 10.3348/kjr.2010.11.1.84. Epub 2009 Dec 28. PMID 20046499
- [Background] Rykkje A, Carlsen JF, Nielsen MB. Hand-Held Ultrasound Devices Compared with High-End Ultrasound Systems: A Systematic Review. Diagnostics (Basel). 2019 Jun 15;9(2):61. doi: 10.3390/diagnostics9020061. PMID 31208078
- [Background] Pudas T, Hurme T, Mattila K, Svedstrom E. Magnetic resonance imaging in pediatric elbow fractures. Acta Radiol. 2005 Oct;46(6):636-44. doi: 10.1080/02841850510021643. PMID 16334848
- [Background] Skaggs DL, Mirzayan R. The posterior fat pad sign in association with occult fracture of the elbow in children. J Bone Joint Surg Am. 1999 Oct;81(10):1429-33. doi: 10.2106/00004623-199910000-00007. PMID 10535592
- [Background] Supakul N, Hicks RA, Caltoum CB, Karmazyn B. Distal humeral epiphyseal separation in young children: an often-missed fracture-radiographic signs and ultrasound confirmatory diagnosis. AJR Am J Roentgenol. 2015 Feb;204(2):W192-8. doi: 10.2214/AJR.14.12788. PMID 25615780
- [Background] Tokarski J, Avner JR, Rabiner JE. Reduction of Radiography with Point-of-Care Elbow Ultrasonography for Elbow Trauma in Children. J Pediatr. 2018 Jul;198:214-219.e2. doi: 10.1016/j.jpeds.2018.02.072. Epub 2018 Apr 19. PMID 29681446
- [Background] Zuazo I, Bonnefoy O, Tauzin C, Borocco A, Lippa A, Legrand M, Chateil JF. Acute elbow trauma in children: role of ultrasonography. Pediatr Radiol. 2008 Sep;38(9):982-8. doi: 10.1007/s00247-008-0935-5. Epub 2008 Jul 15. PMID 18626636
- [Background] Weinberg ER, Tunik MG, Tsung JW. Accuracy of clinician-performed point-of-care ultrasound for the diagnosis of fractures in children and young adults. Injury. 2010 Aug;41(8):862-8. doi: 10.1016/j.injury.2010.04.020. Epub 2010 May 13. PMID 20466368
- [Background] Griffith JF, Roebuck DJ, Cheng JC, Chan YL, Rainer TH, Ng BK, Metreweli C. Acute elbow trauma in children: spectrum of injury revealed by MR imaging not apparent on radiographs. AJR Am J Roentgenol. 2001 Jan;176(1):53-60. doi: 10.2214/ajr.176.1.1760053. PMID 11133538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled through a single emergency room from January 2022 through April 2023.
Pre-assignment Details: This study did not involved randomization. Patient were not randomized for this study. For both feasibility (N=22) and active (N=13) parts of this study, all participants who met inclusion criteria were enrolled. There was no crossover of participants of the two distinct parts of this study.
Units Other Than Participants: Images
Groups:
- Ultrasound Exam: The Study consisted of two parts, a feasibility part and an active part.
  Participants in the feasibility part of the study only underwent a pocket-sized ultrasound exam and were a distinct (unique) group with no overlap or involvement with the active part. Each participant had 10 US images obtained.
  Participants in the active part of the study underwent a pocket-sized ultrasound exam and continued with normal clinically indicated medical care in the ED. The comparison to the ultrasound images was either a X-ray if fracture was suspected or bedside nursemaid reduction if subluxation was suspected (participants acted as their own comparison based on their routine ED clinical management). There was no participation overlap with the feasibility part. Each participant had 10 US images obtained.
Period: Feasibility
Arm/Group | Ultrasound Exam
Started | 22; 440 Images (This was a single group study and there were no separate groups for the feasibility study. All participants enrolled during feasibility had an elbow exam completed and was one time encounter. Participants in feasibility study were not involvement in the active study.)
Completed | 22; 440 Images
Not Completed | 0; 0 Images
Period: Active
Arm/Group | Ultrasound Exam
Started | 13; 260 Images (This was a single group study and there were no separate groups for the active study. All participants enrolled during active had an elbow exam completed and was one time encounter. Participants in active were study not involvement in the feasibility study.)
Completed | 13; 260 Images
Not Completed | 0; 0 Images

BASELINE CHARACTERISTICS:
Groups:
- Ultrasound Exam/Feasibility: Every participant will undergo a pocket-sized ultrasound exam. Both elbows were imaged. Age, gender, and race/ethnicity were not obtained or recorded.
- Ultrasound Exam/Active: Every participant will undergo a pocket-sized ultrasound exam. The comparison to these images either a X-ray if fracture was suspected or beside nursemaid reduction if radial subluxation was suspected (participants acted as their own comparison based on their routine ED clinical management). Race/ethnicity were not obtained or recorded.
- Total: Total of all reporting groups
Arm/Group | Ultrasound Exam/Feasibility | Ultrasound Exam/Active | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 13 | 35
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Mean (Full Range); unit: years] — Patients were screened for age but age was only recorded for the ACTIVE component of this study. It was not collected for the feasibility part (there was also no crossover from the feasibility part of the study to the active part). Population: Age of each participant was not obtained for feasibility part of study.
  years
    Age, Continuous Mean (Full Range): number analyzed (Participants) | 0 | 13 | 13
    Age, Continuous Mean (Full Range) |  | 7 [1 to 14] | 7 [1 to 14]
Sex/Gender, Customized [Number; unit: participants] — Sex/gender was only obtained for the ACTIVE component of this study. It was not collected for the feasibility part (there was also no crossover from the feasibility part of the study to the active part). Population: Gender was not obtained for the feasibility part of the study.
  participants
    Sex/Gender Female (ACTIVE ONLY): number analyzed (Participants) | 0 | 13 | 13
    Sex/Gender Female (ACTIVE ONLY) |  | 9 | 9
    Sex/Gender Male (ACTIVE ONLY): number analyzed (Participants) | 0 | 13 | 13
    Sex/Gender Male (ACTIVE ONLY) |  | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pocket Sized Ultrasound Elbow Exam Interpretation of Fracture
Description: FOR THE ACTIVE STUDY ONLY: Pocket-size ultrasound exam for each participant were interpreted as positive, negative or equivocal for signs of fracture. The feasibility study was not assessing for the presence or absence of fracture.
Time Frame: 1ED visit (1 day)
Population: FOR THE ACTIVE STUDY ONLY: Images will be categorized as positive, negative or equivocal for signs of fracture. Pocket-sized US interpretation was compared to X-ray or performance of bedside nursemaid reduction as gold standard comparison.
  The feasibility study was not assessing for the presence or absence of fracture and did not have data analyzed for this outcome of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Ultrasound Exam/Feasibility: Every participant will undergo a pocket-sized ultrasound exam. Both elbows were imaged.
Arm/Group | Ultrasound Exam/Feasibility | Ultrasound Exam/Active
Number analyzed (Participants) | 0 | 13
Participants
  Pocket-sized US interpretation: Positive Fracture at ED visit on US |  | 8
  Pocket-sized US interpretation: Negative Fracture at ED visit on US |  | 5
  X-ray or Nursemaid Reduction Outcome (Nursemaid reduction considered negative for fracture): Positive Fracture at ED visit on US |  | 7
  X-ray or Nursemaid Reduction Outcome (Nursemaid reduction considered negative for fracture): Negative Fracture at ED visit on US |  | 6
Statistical Analysis 1: Comparison: Ultrasound Exam/Active; Test type: Other — Sample size too small to perform additional statistical tests; Sample size too small to perform additional statistical tests

2. Secondary Outcome: Ultrasound Exam Image Quality
Description: Each participant in both the feasibility and active parts of the study underwent a pocket sized ultrasound exam. 10 ultrasound images were obtained of each elbow and both elbows were imaged. Images will deemed adequate or inadequate for interpretation.
Time Frame: Time period to complete since ultrasound exam per participant, approximately < 15 min
Population: In each part of the study, participants were enrolled and both elbows were imaged, with ten views of each elbow, resulting in 20 images per participant. As result the feasibility study had 440 images reviewed and the active study had 260 images.
Measure: Number; unit: Images
Units Other Than Participants: Images
Arm/Group | Ultrasound Exam/Feasibility | Ultrasound Exam/Active
Number analyzed (Participants) | 22 | 13
Number analyzed (Images) | 440 | 260
Images
  Adequate Image Quality | 413 | 258
  Inadequate Image Quality | 27 | 2
Statistical Analysis 1: Comparison: Ultrasound Exam/Active; Test type: Other — Sample size too small to perform additional statistical tests; Sample size too small to perform additional statistical tests

ADVERSE EVENTS:
Time Frame: 1 ED visit (single day).
Groups:
- Ultrasound Exam/Feasibility; Ultrasound Exam/Active: Every participant will undergo a pocket-sized ultrasound exam of each elbow.
Arm/Group | Ultrasound Exam/Feasibility | Ultrasound Exam/Active
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/13
Other Adverse Events (participants affected / at risk) | 0/22 | 0/13

LIMITATIONS AND CAVEATS:
Given time restraints of the study, slow recruitment and pandemic-related fluctuations in pediatric ED visits, the active portion of the study was not successful in enrolling the sample goal of 70. As a result, the sample size was too small to perform additional statistical tests given poor power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT05870345/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT05870345/ICF_001.pdf